CLINICAL TRIAL: NCT00678574
Title: The Role of GABA and Neurosteroids in Premenstrual Dysphoric Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9803010098
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2017-07

CONDITIONS: Premenstrual Dysphoric Disorder; Premenstrual Syndrome
Keywords: hormones; menses; PMS; PMDD
MeSH Terms: conditions — Premenstrual Dysphoric Disorder; Premenstrual Syndrome | interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Premenstrual Dysphoric Disorder (PMDD) group (Experimental): PMDD group received fluoxetine 20 mg daily by mouth for 2-3 months
  Interventions: Drug: fluoxetine
- Healthy controls (No Intervention)

INTERVENTIONS:
Drug: fluoxetine — Fluoxetine 20 mg daily by mouth for 2-3 months.
  Other Names: Prozac; Sarafem
  Arms: Premenstrual Dysphoric Disorder (PMDD) group

SUMMARY:
The purpose of the study proposed is to investigate the role of neurosteroids and GABA in the pathophysiology and treatment of premenstrual dysphoric disorder (PMDD) by 1) measuring cortical gama-aminobutyric acid levels (GABA levels) using nuclear magnetic resonance spectroscopy (MRS) during the follicular and mid-luteal phases of the menstrual cycle pre and post treatment with the selective serotonin reuptake inhibitor (SSRI) fluoxetine (Prozac®, Sarafem®), and 2) correlating cerebrospinal fluid (CSF) and plasma GABA and neurosteroid levels with cortical GABA levels at these same time points. Neurosteroids to be measured include allopregnanolone, pregnenolone, and pregnenolone sulfate. Findings from women with PMDD will be compared to those of healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 45 years old and able to give voluntary written informed consent.
* Willing to complete a daily log of mood symptoms for 7 consecutive menstrual cycles: two menstrual cycles during the Screening Phase (Phase 1), one menstrual cycle during the Testing Phase (Phase 2), and four menstrual cycles during the Medication Treatment Phase and Post-Treatment Phase (Phase 3). All subjects who successfully complete Phases 1 and 2, and the Medication Treatment Phase, will be invited to participate in Phase 3 approximately three months later. Phase 3 will involve repeating all procedures conducted in Phase 2, including the daily log of mood symptoms.
* Meet DSM-IV criteria for premenstrual dysphoric disorder, confirmed by the Daily Record of Severity of Problems (DRSP; Endicott & Harrison) for 2 consecutive menstrual cycles (Phase 1). The DRSP is a self-rated symptom checklist, which requires individuals to rate their symptoms of PMDD according to the DSM-IV research criteria scale on a scale from 1 (symptom not present) to 6 (symptom extreme). During the last 7 days of the menstrual cycle compared to days 5-11, patients must have a 30% increase in their average (over 2 menstrual cycles) score for 5 of these 10 symptoms. Symptoms must be "not present" or "minimal" during the postmenstrual week.
* Average 19-item Hamilton Depression Rating Scale (HAM-D) scores < 5 during the follicular phase and > 16 during the luteal phase.
* Have regular menstrual cycles 28 to 32 days in length. Each of the screening cycles must be ovulatory as confirmed by plasma progesterone levels of >5 ng/ml during the luteal phase.

Exclusion Criteria:

* Presence of any other comorbid DSM-IV Axis I disorder.
* Meeting DSM-IV criteria for psychoactive substance (excluding nicotine) dependence within the preceding 4 months.
* A history of serious medical or neurological illness, including (but not limited to) major cardiovascular disease, severe hypertension, intracranial mass lesions, seizure disorder, severe hepatic or renal disease, unstable endocrine or metabolic disease, and unstable hematologic disease.
* Use of anticonvulsant or benzodiazepines within the last month.
* Use of psychotropic medication in last week (except as stated above).
* Use of steroid contraceptives within the previous 4 months, including birth control pill, birth control patch, birth control ring, and Depo-Provera®. Subjects will be asked to use abstinence or the barrier method (condoms) as forms of contraception in this study.
* Alcohol consumption greater than 7 drinks/week.
* Current pregnancy.
* Metallic implants.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 1998-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, MD, Principal Investigator — University of Pennsylvania School of Medicine Department of Psychiatry
Locations (1):
- Yale University, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 subjects were recruited at an outpatient practice at Yale University, CT.
Groups:
- PMDD: Participants who qualified as having PMDD received fluoxetine 20 mg daily by mouth for 2-3 months
- Healthy Controls: Participants who did not qualify for a diagnosis of PMDD and did not receive drug treatment.
Period: Overall Study
Arm/Group | PMDD | Healthy Controls
Started | 18 | 27
Completed | 18 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PMDD Group: Fluoxetine 20 mg daily by mouth for 2-3 months to the PMDD group
- Healthy Controls: No intervention was provided to the healthy control group.
- Total: Total of all reporting groups
Arm/Group | PMDD Group | Healthy Controls | Total
Number analyzed (Participants) | 18 | 27 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 27 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Cortical Gama-aminobutyric Acid Levels (GABA Levels) Pre and Post SSRI Treatment
Description: GABA levels would be assessed during the follicular and mid-luteal phases of the menstrual cycle pre and post treatment with the SSRI.
Time Frame: 2-3 months post-treatment w/ fluoxetine.
Population: This study was conducted at Yale several years ago. Our group at UPenn only has basic information about this study. This includes the number of participants, which was 18, and that no adverse events occurred. The contact person who initially entered this study protocol information is no longer at the University of Pennsylvania.
Groups:
- Fluoxetine: Fluoxetine 20 mg daily by mouth for 2-3 months in PMDD group
- No Intervention: No intervention was provided in the healthy control group.
Arm/Group | Fluoxetine | No Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the course of the study.
Groups:
- No Treatment: Healthy controls received no treatment.
Arm/Group | Fluoxetine | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/27
Other Adverse Events (participants affected / at risk) | 0/18 | 0/27

LIMITATIONS AND CAVEATS:
Data from this study has not yet been analyzed nor peer reviewed. As much information as possible was entered into the results section of this trial, however information is missing as it pertains to specific measurements collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes